CLINICAL TRIAL: NCT06724263
Title: A Multicenter, Open-label Phase IIa Clinical Study to Evaluate the Efficacy and Safety of B1962 Injection in the Treatment of Advanced Malignant Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Biopharmaceuticals Co., Ltd. (Industry)
Collaborators: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSL-B1962-02
Record Dates: First submitted 2024-11-28; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Platinum-resistant Epithelial Ovarian Cancer; Triple Negative Breast Cancer (TNBC); Cervical Cancers; Small Cell Lung Cancer; Hepatocellular Carcinoma (HCC); Colorectal Cancer; Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Uterine Cervical Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Hepatocellular; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B1962 (Experimental): advanced malignant neoplasm
  Interventions: Drug: B1962

INTERVENTIONS:
Drug: B1962 — B1962 has higher VEGF anti angiogenic activity than its competitors. Phase I clinical trials have shown that B1962 has excellent safety and promising therapeutic effects. Large scale clinical studies may achieve better therapeutic effects than similar competitors targeting the same target
  Other Names: B1962 is a PD-L1/VEGF bispecific antibody fusion protein.

SUMMARY:
This is a multicenter, open-label Phase IIa clinical study to evaluate the efficacy and safety of B1962 in the treatment of ad-vanced solid tumors.

The study consists of a Screening Period, a Treatment Period, and a Follow-up Period (EOT Visit, Safety Follow-up, and Survival Follow-up).

Subjects who meet the inclusion criteria and do not meet the exclusion criteria at screening will enter the appropriate study co-hort according to tumor type and receive B1962 until unacceptable toxicity, radiographic disease progression, or withdrawal of the sub-ject for other reasons, whichever comes first, for a maximum of 24 months of treatment. Enrollment will be conducted according to three stages: Stage I: It is planned to enroll 5 patients in each of 8 cohorts (tumor type) to observe the safety and efficacy; Stage II: 1 ~ 2 cohorts are preferred to enroll 15 ~ 20 patients to observe the ef-ficacy and safety; Stage III: 1 cohort is finally preferred to continue enrollment until a total of no more than 60 patients are observed in this cohort to observe the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be eligible for enrollment in this study:

  1. Voluntary participation in the study and provision of signed and dated informed consent;
  2. Age ≥ 18 years at the time of informed consent;
  3. Patients with histologically or cytologically confirmed advanced malignant solid tumors who have failed or failed to respond to first-line standard therapy, or cannot tolerate standard therapy, or have no standard effective treatment regimen, or refuse standard therapy; and no more than 4 lines of prior systemic anti-tumor therapy. Specific tumor species cohorts were as follows:

     * Recurrent platinum-resistant epithelial ovarian cancer (including primary peritoneal and/or fallopian tube cancer): pathologically confirmed ovarian epithelial malignancy, fallopian tube epithelial malignancy, primary peritoneal cancer; and diagnosed platinum-resistant (duration of response to platinum-based therapy is within 6 months after the last dose of platinum-based therapy)

       * Triple-negative breast cancer: pathologically confirmed unresectable locally advanced or metastatic breast cancer with negative ER, PR, and HER-2. ER, PR negativity was defined as: IHC ER < 1%, IHC PR < 1%. HER-2 negativity is defined as IHC HER-2 (-) or (1 +), and FISH must be performed and the result is negative for HER-2 (2 +) ③ Cervical cancer: pathologically confirmed inoperable locally advanced or metastatic cervical cancer

         * Small-cell lung cancer: histologically or cytologically confirmed, inoperable, locally advanced or metastatic small-cell lung cancer

           ⑤ Biliary Tract Cancer: Pathologically confirmed unresectable locally advanced or metastatic biliary tract cancer, including gallbladder cancer and intrahepatic and extrahepatic cholangiocarcinoma

           ⑥ Hepatocellular carcinoma: pathologically confirmed hepatocellular carcinoma (excluding mixed hepatocellular carcinoma); Barcelona Clinic Liver Cancer (BCLC) stage C, not suitable for radical surgery and/or local treatment or stage B without radical progression after surgery and/or local treatment; Child-Pugh A liver function; for patients with esophagogastric varices, if gastroscopy or imaging, ultrasound and other examinations suggest severe (G3) varices or positive red sign, indicating high risk of venous bleeding, they are not allowed to participate in this study.

           ⑦ Colorectal cancer: pathologically confirmed unresectable locally advanced or metastatic colorectal cancer

           ⑧ Non-squamous non-small cell lung cancer: pathologically confirmed unresectable locally advanced or metastatic non-squamous non-small cell lung cancer that cannot contain a small cell lung cancer component.
  4. Willingness to comply with protocol-specified visits, study treatment, laboratory tests, and other study-related procedures and requirements;
  5. Eastern Cooperative Oncology Group (ECOG) performance score 0-1;
  6. Expected survival time of more than 3 months;
  7. Presence of at least one measurable lesion (non radiation therapy field) confirmed by CT or MRI that meets RECIST v1.1 criteria;
  8. Adequate organ and bone marrow function:

     Hematologic system (no transfusion, no G-CSF use, no medication for correction within 2 weeks prior to screening): absolute neutrophil count (ANC) ≥ 1.5 × 10 9/L, platelets (PLT) ≥ 75 × 10 9/L, hemoglobin (Hb) ≥ 90 g/L； Liver function: total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 3.0 × ULN, aspartate aminotransferase (AST) ≤ 3.0 × ULN; for patients with liver metastasis: ALT ≤ 5.0 × ULN, AST ≤ 5.0 × ULN;

     Renal function:

     i. Creatinine ≤ 1.5 × ULN, or creatinine clearance (Ccr) ≥ 50 mL/min (calculated according to Cockcroft-Gault formula *);

     * Formula is: Ccr (ml/min) = [(140-age) × weight kg × F]/[serum creatinine (mg/dl) × 72] (F = 1 for males and 0.85 for females) ii. Urine protein < 2 + (ie, 0, ± or 1 +) or proteinuria ≤ 1 g/24 hours Note: All patients with ≥ 2 + urine protein in urinalysis must have a 24-hour urine collection and proteinuria ≤ 1 g/24 hours must be confirmed Coagulation: prothrombin time (PT) ≤ 1.5 × ULN or international normalized ratio (INR) ≤ 1.5 × ULN, and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
  9. For female patients:

     Females of childbearing potential, who are not breastfeeding, agree to use highly effective contraception from signing the ICF and use this contraception during the study and for 3 months after the last dose; blood pregnancy results (human chorionic gonadotropin hCG) must be negative within 7 days prior to enrollment; Females of non-childbearing potential (ie, physiologically incapable of becoming pregnant), including those surgically sterilized (having undergone bilateral oophorectomy, bilateral tubal ligation, or hysterectomy), or postmenopausal for ≥ 12 months prior to Screening (amenorrhea not due to treatment);
  10. Male patients with female partners of childbearing potential must agree to use highly effective contraception starting from signing the ICF and for the duration of the study and for 3 months after the last dose.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from the study:

  1. Prior use of anti-PD-1 monoclonal antibody, anti-PD-L1 monoclonal antibody, or other antineoplastic agents containing PD- (L) 1 target;
  2. Patients who have previously used macromolecular VEGF/VEGFR inhibitors such as bevacizumab, ramucirumab;
  3. Known hypersensitivity to the study drug or any of its components, or previous severe hypersensitivity to macromolecular protein preparations/monoclonal antibodies or bispecific antibodies;
  4. Female patients are pregnant or lactating;
  5. Major surgery within 4 weeks prior to the first dose of study drug, or planned major surgery within the study period; For primary or metastatic liver cancer: local treatment of liver (such as transarterial chemoembolization, transcatheter embolization, hepatic arterial infusion, radiotherapy, radioembolization or radiofrequency ablation, etc.) within 4 weeks prior to the first dose of study drug;
  6. Adverse reactions from prior anticancer therapy that have not recovered to NCI-CTCAE v5.0 grade ≤ 1 (except alopecia and other for which the investigator considers there is no safety risk);
  7. Patients with clinical symptoms of brain metastases, spinal cord compression, carcinomatous meningitis, or patients with other evidence of uncontrolled brain or spinal cord metastases (except for stable symptoms and imaging studies showing stable disease for at least 4 weeks before the first dose);
  8. Patients with clinical symptoms or pleural effusion, pericardial effusion or ascites requiring repeated drainage;
  9. Screening imaging showed tumor encasing vital blood vessels or obvious necrosis and cavity, and the investigator judged that entering the study would cause bleeding risk; according to anatomical classification of tumor location, diagnosis of central lung cancer, or tumor involving hilum with bleeding risk.
  10. Known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive) or acquired immunodeficiency syndrome-related disease;
  11. Positive hepatitis B surface antigen (HBsAg), and HBV DNA higher than the upper limit of normal value of the detection unit; or positive hepatitis C antibody (HCV-Ab) and HCV-RNA quantification > the upper limit of normal value of the detection unit; or known active syphilis infection;
  12. Uncontrolled bacterial, viral, fungal infections and other pathogen infections (such as mycoplasma, parasites, etc.) requiring systemic treatment within 4 weeks prior to the first dose of study drug;
  13. History of significant cardiovascular disease, including but not limited to: malignant arrhythmia requiring clinical intervention; or acute coronary syndrome (myocardial infarction and angina pectoris) within 6 months prior to the first dose; or congestive heart failure meeting New York Heart Association (NYHA) functional class II or higher criteria; or left ventricular ejection fraction (LVEF) < 50%; poorly controlled hypertension with standard treatment or poor compliance with antihypertensive therapy; history of hypertensive crisis or hypertensive encephalopathy; and significant vascular disease (eg, aortic aneurysm requiring surgery);
  14. Patients with coagulation disorders, bleeding disorders, or other conditions judged by the investigator to be at risk of bleeding, such as skin wounds, surgical sites, wound sites, severe mucosal ulcers or fractures that have not healed completely, or active gastroduodenal ulcers, gastrointestinal bleeding, intestinal obstruction, ulcerative colitis, esophagogastric varices, gastrointestinal perforation within 6 months prior to the first dose;
  15. Pulmonary hemorrhage/hemoptysis (daily bleeding/hemoptysis volume ≥ 2.5ml) within 4 weeks prior to the first dose of study drug;
  16. Biopsy or other minor surgery within 7 days prior to the first dose of study drug, excluding placement of vascular access devices;
  17. Arterial or venous thrombosis, or stroke or transient ischemic attack within 6 months prior to the first dose of study drug;
  18. Unstable anticoagulant or thrombolytic therapy within 14 days of the first dose of study drug;
  19. Chronic treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory drugs known to inhibit platelet function, or thienopyridines such as ticlopidine, clopidogrel, or phosphodiesterase inhibitors such as dipyridamole, cilostazol within 14 days of the first dose of study drug;
  20. Diabetes mellitus not stably controlled by drug therapy; thyroid diseases not stably controlled by drug therapy, such as hyperthyroidism;
  21. Current or previous idiopathic pulmonary fibrosis or idiopathic pneumonia; current acute lung disease, interstitial lung disease or pneumonia (except for local interstitial pneumonia induced by radiotherapy), pulmonary fibrosis, etc.; severe dyspnea, pulmonary insufficiency or continuous oxygen inhalation for any reason;
  22. Active autoimmune diseases or history of autoimmune diseases requiring systemic treatment within 2 years before screening, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis or glomerulonephritis; Exceptions: hypothyroidism controlled by hormone replacement therapy alone, dermatologic conditions not requiring systemic therapy (eg, vitiligo, psoriasis), controlled celiac disease;
  23. Systemic corticosteroid therapy (prednisone > 10 mg/day or equivalent of the same class) or systemic therapy with other immunosuppressive agents within 14 days prior to the first dose of study drug; Exceptions include treatment with topical, ocular, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption, or prophylactic short-term (≤ 7 days) use of corticosteroids (eg, allergy to contrast agents), or for the treatment of non-autoimmune conditions (eg, delayed hypersensitivity caused by contact allergens);
  24. Received the last systemic anti-tumor therapy (biological agent therapy, etc.) within 4 weeks prior to the first dose, chemotherapy or hormone anti-tumor therapy within 2 weeks prior to the first dose, received non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, cyclophosphamide, methotrexate, thalidomide, tumor necrosis factor, etc.) within 2 weeks prior to the first dose, and received Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 1 week prior to the first dose ;
  25. Prior organ or hematopoietic stem cell transplant;
  26. History of other neoplasms within 5 years prior to screening, except cured cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma, who had undergone successful radical surgery;
  27. Has received attenuated vaccines within 4 weeks prior to Screening or plans to receive attenuated vaccines during the study;
  28. Patients who participated in a clinical study and received study drug within 4 weeks prior to the first dose;
  29. History of alcohol or drug abuse within 12 months prior to the first dose;
  30. Known psychiatric disorder that could affect trial compliance;
  31. Other serious systemic diseases or laboratory abnormalities or other reasons considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  Proportion of patients who achieved complete response (CR) or partial response (PR) at two consecutive reviews ≥ 4 weeks apart.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No